CLINICAL TRIAL: NCT04482361
Title: SERO-EPIDEMIOLOGY OF SARS-COV2 INFECTION IN THE AUTONOMOUS CITY OF BUENOS AIRES
Status: Completed | Type: Observational
Sponsor: Ministerio de Salud de Ciudad Autónoma de Buenos Aires (Other Government)
Responsible Party: Sponsor
Other Study IDs: SEROEPIDEMIOLOGY COVID IN CABA
Record Dates: First submitted 2020-07-20; First posted 2020-07-22 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: COVID-19
Keywords: Seroepidemiology; Epidemiology; Antibodies
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Presence of specific anti-SARS-CoV-2 antibodies — Presence of specific anti-SARS-CoV-2 antibodies

SUMMARY:
The pandemic of a new coronavirus SARS-COV-2, which causes COVID-19 disease, has spread rapidly and is a major public health challenge. While the focus is primarily on containing the number of cases and finding alternative therapies, information is still lacking to elucidate the dynamics of viral circulation and to understand the distribution of the infection in the population.

The cases reported in Argentina and worldwide could plausibly represent only a small proportion of the number of asymptomatic or poorly symptomatic cases that exist in society. However, the magnitude of this dissociation between symptomatic cases and asymptomatic persons is unknown.

Knowing this information is of strategic importance as it will allow the estimation of a community prevalence and the evaluation of the best containment strategy. In fact, although all social distancing measures are now indispensable, the feasibility of prolonging the measure over time is a complex issue and in any case will require population-based information.

The best way to approach the estimation of a true population prevalence is to take representative samples from the population and test them periodically. These experiences were carried out in other contexts showing heterogeneous results within the community studied. In Spain, for example, the range of antibodies present in the population varied from 1.1% to 14.2%, also showing that an important part of the population had had contact with the virus without symptoms. Studies in Switzerland and the United States also show similar findings. However, these estimates are not automatically transferable to other settings.

The city of Buenos Aires has a particular demographic composition with an important group of the population living in shantytowns (it is estimated that between 7% and 10% of the population lives in shantytowns) and with much heterogeneity among the different communes of the city. In the villas, the incidence rates of COVID-19 infection differ significantly from those present in the group "outside the village". However, there is also an important difference in the incidence rates by commune, even without considering the villas.

Thus, it is important to know the sero-epidemiology of antibodies against SARS-COV2 in a representative sample of the city of Buenos Aires.

For this purpose, a nationally produced test (COVIDAR IgG) developed by professionals from CONICET and Instituto Leloir will be used.

The aim of this initiative is to estimate the true dimension of the COVID-19 epidemic in the City of Buenos Aires, by studying the immunological status of the Buenos Aires population in relation to SARS-Cov2, as well as to observe the evolution of the infection among the population, since this information is essential to guide future public health measures related to the control of COVID-19.

To achieve this objective, a comprehensive sero-epidemiological study will be carried out to provide estimates of past SARS-Cov2 infection with sufficient precision to be representative of the sero-epidemiological status of the Buenos Aires city population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 at the time of signing the informed consent

Exclusion Criteria:

* ≤17 years old.
* Declare that currently having confirmed COVID-19 infection.
* Inability to give informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The present study will be a transversal study carried out on 1,800 people over 18 years of age resident in CABA for 10 working days, between the months of July and August. The survey will be repeated in August and September.
Sampling Method: Probability Sample
Enrollment: 5900 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2020-12-22 (Actual)

PRIMARY OUTCOMES:
Prevalence of IGG for COVID-19 | 4 months
  To estimate the prevalence of SARS-Cov2 infection in the city of Buenos Aires, by means of the determination of IGG-type antibodies in a representative and randomized sample of adult residents of the city.
Changes in prevalence of IGG for COVID-19 | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ministerio de Salud de la Ciudad Autónoma de Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No